CLINICAL TRIAL: NCT05490979
Title: Effectiveness and Physiological Mechanisms of Contemplative Dyad Meditation to Increase Social Connection in Young Adults in the Aftermath of the Pandemic
Brief Title: The Impact of Dyad Exercises on Well-being and Connection in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Michael Platt, James S. Riepe University Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #10085952
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Mental Health Wellness 1; Loneliness

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants only receive information about the condition they have been assigned to and are not explicitly informed about the other conditions or the overall purpose of the study. All participants will be debriefed when the study has ended.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Contemplative dyad meditation (Experimental)
  Interventions: Behavioral: Contemplative dyad meditation
- Fast friends (Active Comparator)
  Interventions: Behavioral: Fast friends
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Contemplative dyad meditation — Participants take part in a 3-hour group meditation training led by a professional meditation teacher. They receive detailed instructions and also practice contemplative dyad meditation for at least 30 minutes with another participant. During the 2 weeks following the training, participants meet in supervised group settings to practice the meditation method with alternating partners for up to 6 times.
  Arms: Contemplative dyad meditation
Behavioral: Fast friends — During 2 weeks, participants meet in supervised group settings to practice the 'fast friends' exercise with alternating partners for up to 6 times.
  Arms: Fast friends

SUMMARY:
Many people are experiencing low well-being and loneliness, particularly due to the COVID-19 pandemic. As the world is opening back up, it is crucial to determine methods to help people grow closer again and boost subjective well-being. One promising method is contemplative dyad meditation, which has hardly been studied. This is a method in which two people have a structured dialogue with each other while contemplating a prompt, as they alternate between listening and speaking. It is related to but different from other methods that have previously been shown to increase connection, such as the "fast friends" exercise. In "fast friends", two people answer a series of increasingly personal questions in a dialogue.

Here, 180 participants between 18-35 years will be randomly allocated to three conditions (stratified by gender): (a) contemplative dyad meditation training, (b) "fast friends", or (c) no-intervention. Participants in the dyad meditation group will receive professional meditation training followed by 2 weeks of regular meditation practice. Participants in the "fast friends" group will meet regularly during 2 weeks to practice "fast friends" exercises. The impact of the interventions on well-being, loneliness, mindfulness, and related measures will be investigated. After the interventions have finished, participants' physiology (heart rate) and brain waves (using electroencephalography [EEG]) during the respective exercises will also be measured to explore potential biological mechanisms. Of particular interest are heart rate variability (HRV, often linked with higher well-being), frontal alpha asymmetry in the EEG (linked with positive affect and approach), and biological synchrony in these variables between the two interacting individuals.

Both dyad meditations and "fast friends" exercises are predicted to improve closeness, thriving, loneliness, affect, depression, anxiety, and social interaction anxiety compared to no-intervention. Moreover, dyad meditation is predicted to have stronger effects than "fast friends" in terms of increasing mindfulness, self-compassion, and empathy. Dyad meditation and fast friends will show differential physiological signatures (e.g., lower heart rate and higher averaged alpha power for meditation).

This study may reveal effective methods to improve well-being and connection and provide insights into their biological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Current student, staff, or employee at the University of Pennsylvania (for safety reasons)

Exclusion Criteria:

* none

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Brief Inventory of Thriving | 3 weeks
  The Brief Inventory of Thriving (Su, Tay, & Diener, 2014) is a questionnaire consisting of 10 items, measuring psychological well-being. Scores range from 1 to 5 with a higher score indicating more thriving (i.e., higher well-being).
Loneliness Scores on the Comprehensive Inventory of Thriving | 3 weeks
  The Loneliness sub-scale from the Comprehensive Inventory of Thriving (Su, Tay, & Diener, 2014) consists of 3 items. Scores range from 1 to 5 with a higher score indicating higher loneliness.
Mindfulness Score on the Five Facet Mindfulness Questionnaire | 3 weeks
  The Five Facet Mindfulness Questionnaire (Baer et al., 2006) consists of 39 items. Scores for mindfulness range between 1 and 5 with a higher score indicating more mindfulness.
Inclusion of Other in the Self Scale | Directly after each individual meditation or "fast friends" exercise
  The Inclusion of Other in the Self Scale (Aron, Aron, & Smollan, 1992) consists of 7 response options measuring closeness to another person (here: the meditation or exercise partner). The response options each show two circles labeled as" "Self" and "Other", which vary in terms of overlap, from barely touching (1, i.e., not close at all) to almost completely overlapping (7, i.e., extremely close).

SECONDARY OUTCOMES:
Positive Affect Scores on the Negative And Positive Affect Scale | 3 weeks
  The 10-item version of the Negative And Positive Affect Scale by Joshanloo (2017) contains 5 items measuring positive affect. Scores for positive affect from these 5 items range from 5 to 25 with 25 indicating higher positive affect. The scale is used here with the following adaptation: it asks about the previous 14 days rather than 30 days.
Negative Affect Scores on the Negative And Positive Affect Scale | 3 weeks
  The 10-item version of the Negative And Positive Affect Scale (NAPAS) by Joshanloo (2017) contains 5 items measuring negative affect. Scores for negative affect from these 5 items range from 5 to 25 with 25 indicating higher negative affect. The scale is used here with the following adaptation: it asks about the previous 14 days rather than 30 days.
Depression Scores on the Patient Health Questionnaire-9 | 3 weeks
  The Patient Health Questionnaire-9 consists of 9 items and measures the severity of depression. Scores range from 0 to 27 with a higher score indicating more severe depression.
Generalized Anxiety Disorder-7 questionnaire | 3 weeks
  The Generalized Anxiety Disorder 7-item questionnaire screens for general anxiety disorder. Scores range from 0 to 21 with higher scores indicating more severe anxiety.
Social Interaction Anxiety Scale-6 | 3 weeks
  The Social Interaction Anxiety Scale-6 (Peters et al., 2012) is a 6-item measure assessing social interaction anxiety. Scores range from 0 to 24 with 24 indicating more severe social anxiety.
Self-Compassion Scale Short-Form | 3 weeks
  The short form of the Self-Compassion Scale (Raes et al., 2011) includes 12 items. Scores range from 1 to 5 with higher scores indicating more self-compassion. Change = (Week 3 Score - Baseline Score).
Toronto Empathy Questionnaire | 3 weeks
  The Toronto Empathy Questionnaire consists of 16 items. Scores range from 0 to 64 with higher scores indicating higher empathy.
Positive Affect Scores on the Negative And Positive Affect Scale | Directly after each individual meditation or "fast friends" exercise
  The 10-item version of the Negative And Positive Affect Scale by Joshanloo (2017) contains 5 items measuring positive affect. Scores for positive affect from these 5 items range from 5 to 25 with 25 indicating higher positive affect. The scale is used here with the following adaptation: it asks about the current moment rather than the past 30 days. Response options are adapted to vary from 1 (not at all) to 5 (extremely).
Negative Affect Scores on the Negative And Positive Affect Scale | Directly after each individual meditation or "fast friends" exercise
  The 10-item version of the Negative And Positive Affect Scale (NAPAS) by Joshanloo (2017) contains 5 items measuring negative affect. Scores for negative affect from these 5 items range from 5 to 25 with 25 indicating higher negative affect. The scale is used here with the following adaptation: it asks about the current moment rather than the past 30 days. Response options are adapted to vary from 1 (not at all) to 5 (extremely).
Emotional synchrony | Directly after each individual meditation or "fast friends" exercise
  Average correlation between emotions of the 2 people doing the exercise together, as reported with regards to the last 5 minutes of the meditation or the "fast friends" exercise. The following emotions (taken from the short version of the Negative and Positive Affect scale by Joshanloo) will be rated by both participants: restless/fidgety, hopeless, that everything was an effort, in good spirits, calm and peaceful, full of life.

OTHER OUTCOMES:
Heart rate | 3 weeks
  measured using electrocardiogram, by Bitalino
Heart rate variability | 3 weeks
  measured using electrocardiogram, by Bitalino, calculated as Root Mean Square of Successive Differences (RMSSD)
Respiration | 3 weeks
  measured using respiration belts by Bitalino
EEG | 3 weeks
  measured using Emotiv-EEG

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Platt, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States